CLINICAL TRIAL: NCT06023537
Title: Using Technology to Investigate Dietary and Physical Activity Lapses in a Behavioral Weight Loss Program
Brief Title: Using Technology to Investigate Lapses in a Weight Loss Program Among Individuals With Overweight and Obesity
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Williams College (Other)
Collaborators: Temple University (Other)
Responsible Party: Principal Investigator, Rebecca Crochiere, Assistant Professor of Psychology, Williams College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-08
Record Dates: First submitted 2023-08-21; First posted 2023-09-05 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Obesity; Weight Loss
Keywords: Obesity; Weight Loss; Behavioral Treatment; Dietary Lapse; Physical Activity Lapse
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral Weight Loss Intervention (Experimental)
  Interventions: Behavioral: Behavioral weight loss program

INTERVENTIONS:
Behavioral: Behavioral weight loss program — All participants will participate in the same remote, behavioral weight loss program. As part of the baseline assessment, participants will be asked to watch a series of custom-made videos on the study's dietary and physical activity prescriptions, dietary self-monitoring, self-weighing, and cognitive-behavioral skills to facilitate engagement in study prescriptions. Participants will be prescribed a reduced-calorie diet that will be individualized based on the individual's starting weight and weight loss goal (recommended goal of 5-10% weight loss over 12 weeks). Participants also will be prescribed a goal of 150 minutes of moderate-to-vigorous physical activity per week. They are also given, free of cost, a Fitbit Charge 5 health tracker, the Fitbit Aria Air digital scale, and a MyFitnessPal Premium subscription for the duration of the study.

SUMMARY:
Approximately 70% of American adults have overweight/obesity, which increases risk of major medical issues and preventable death (Abdelaal et. al, 2017). Many individuals with overweight/obesity attempt to lose weight through behavioral strategies, e.g., adopting a reduced-calorie diet and/or increased physical activity. However, it is exceedingly difficult to consistently adhere to a reduced-calorie diet and high levels of physical activity; as such, most individuals attempting to lose weight via these methods experience repeated instances of non-adherence, i.e., dietary and physical activity lapses. These lapses are a core driver of weight loss failure, undermining individuals' ability to achieve weight control (Forman et al, 2017). As such, it is important to understand what predicts these lapses, which in turn allows for better lapse prevention. The current study proposes to measure these risk factors in an ecologically valid manner, i.e., in the moment they occur and in the context of individuals' everyday lives, using advanced technology. Specifically, the current study will use ecological momentary assessments (EMA; brief, repeated surveys delivered in one's natural environment, typically via a smartphone) and sensor technology (e.g., Fitbit and sensors on smartphone devices) to measure momentary risk factors of dietary and physical activity lapse, as well as the lapses themselves. Findings from this research project will lay the groundwork for a sophisticated just-in-time adaptive intervention (JITAI), a tailored, personalized intervention that targets momentary risk factors (e.g., cravings) via in-the-moment support, thereby reducing lapse occurrence and improving adherence to behavioral weight control prescriptions.

ELIGIBILITY:
Inclusion Criteria:

* Current BMI = 27-50 kg/m2
* Adult (aged 18-65)
* Lives in the United States
* Possession of a smartphone with a data plan that allows for app data collection
* Ability to understand and provide informed consent
* Proficiency in speaking, reading, and writing English

Exclusion Criteria:

* Presently involved in another weight loss program
* Currently pregnant or plan to become pregnant within the study period
* Have a medical condition or psychiatric symptoms that: may pose a risk to the participant during the program; cause a change in weight, appetite, or eating behavior; or limit ability to comply with the program
* Endorse eating disordered behavior, including loss of control (LOC) eating, or the subjective experience that one cannot control how much food he or she consumes
* Have experienced a recent (i.e., within the last 3 months) change in a weight-influencing medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2025-08-14 (Estimated); Study Completion 2025-08-14 (Estimated)

PRIMARY OUTCOMES:
Physical activity lapse/intention-behavior gap | up to 12 weeks
  Physical activity lapse/intention-behavior gap will be measured using ecological momentary assessment (EMA; brief, smartphone-delivered surveys) and accelerometers. EMA surveys will be delivered in 2-week bursts at the beginning, middle, and end of treatment. There will be 6 EMA surveys delivered every 2-3 hours throughout the day. Each EMA survey will ask about the participant's intention to engage in moderate-to-vigorous physical activity (MVPA) in the next 2-3 hours and actual engagement in MVPA. Actual MVPA also will be measured through accelerometers (Fitbits). Thus, by measuring intention to engage in MVPA in the next 2-3 hours at Time 1 (e.g., EMA survey at 9:00am) and if the participant actually engaged in MVPA via accelerometer and EMA at Time 2 (2-3 hours later, e.g., at 12:00pm), we can detect a physical activity intention-behavior gap or physical activity lapse.

SECONDARY OUTCOMES:
Dietary lapse | up to 12 weeks
  A dietary lapse will be operationalized as exceeding an individualized calorie target for a meal/snack. Specifically, participants will be assigned a reduced-calorie diet to facilitate weight control and each will be prescribed a personalized daily calorie target. That target will then be divvied up into individual calorie targets for 3 meals and 2 snacks daily (e.g., 15% of daily calorie goal allotted for breakfast, 25% for lunch, 40% for dinner, and 10% for each of two snacks). If a participant exceeds one of these meal-specific calorie targets, it is considered a dietary lapse. Participants will log everything they eat and drink in MyFitnessPal, which automatically calculates calories and stores participant's calorie goals for meals/snacks; thus, lapses can be identified when a participant exceeds a calorie target for a meal/snack in MyFitnessPal. Participants also will report dietary lapses via EMA surveys (see above for more information about EMA surveys).

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca J Crochiere, PhD, Principal Investigator — Williams College
Locations (1):
- Health Lab, Psychology Department, Williams College, Williamstown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data and analytic code from this study are available (as allowable according to Institutional Review Board standards) upon reasonable request by emailing the principal investigator.